CLINICAL TRIAL: NCT04351880
Title: Meals MATTER: A Randomized Controlled Trial of Medically Tailored Meals 2 Weeks vs. 4 Weeks Post Hospital Discharge
Brief Title: Meals MATTER: A Trial of Medically Tailored Meals 2 Weeks vs. 4 Weeks Post Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-1556587
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure; Copd; Liver Failure; Diabetes Mellitus; Cancer; End Stage Renal Disease
Keywords: medically tailored meals; chronic conditions; food service
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Liver Failure; Diabetes Mellitus; Neoplasms; Kidney Failure, Chronic; Chronic Disease

STUDY DESIGN:
Intervention Model Description: This is a randomized trial to compare two approaches to meal delivery. Group 1 will receive meal delivery for 2 weeks (1 meal per day for a total of 14 days) and Group 2 will receive meal delivery for 4 weeks (1 meal per day for a total of 28 days). A concurrent propensity matched control group which will not receive an intervention will also be used.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meals - 2 weeks (Active Comparator): Receive meal delivery for 2 weeks (1 meal per day for a total of 14 days). The medically tailored meal ordered for each participant will depend on their medical conditions.
  Interventions: Other: Medically Tailored Meals
- Meals - 4 weeks (Active Comparator): Receive meal delivery for 4 weeks (1 meal per day for a total of 28 days). The medically tailored meal ordered for each participant will depend on their medical conditions.
  Interventions: Other: Medically Tailored Meals

INTERVENTIONS:
Other: Medically Tailored Meals — Compare 2 and 4 weeks of meal delivery

SUMMARY:
The purpose of this study is to determine if medically tailored meals provided for either 2 weeks or 4 weeks (1 meal per day) to a Kaiser Permanente Colorado (KPCO) member after hospital discharge will improve their health. Medically tailored meals (MTM) are meals that are approved by a dietitian and shown to help people with certain health conditions.

DETAILED DESCRIPTION:
The purpose of this study is to determine if medically tailored meals provided for either 2 weeks or 4 weeks (1 meal per day) to a Kaiser Permanente Colorado (KPCO) member after hospital discharge will improve their health. Medically tailored meals (MTM) are meals that are approved by a dietitian and shown to help people with certain health conditions.

The Investigators propose a research study with four Specific Aims:

Specific Aim 1: To determine if MTM provided post hospitalization for 4 weeks to patients with one or more of seven chronic health conditions will decrease depression/anxiety measured by the Hospital Anxiety and Depression Scale (HADS) at 60 days in comparison to meals provided for 2 weeks to members discharged from two hospitals.

Hypothesis 1: Patients receiving meals for 4 weeks will have a clinically significant increase in their HADS score at 60 days compared to those receiving meals for 2 weeks.

Specific Aim 2: To determine if MTM provided for 4 weeks to patients with one or more of seven chronic health conditions post hospitalization will improve general well-being and functional status measured by Katz's Activities of Daily Living (ADL).

Hypothesis 2: Patients receiving meals for 4 weeks will have a clinically significant increase in their sense of well-being and ADLs at 60 days compared to those receiving meals for 2 weeks.

Specific Aim 3: To determine if MTM provided for 4 weeks to patients with one or more of seven chronic health conditions post hospitalization will decrease a composite outcome of rehospitalizations and emergency department (ED) visits at 60 days in comparison to: a) meals provided for 2 weeks to members discharged from two hospitals; and b) a concurrent prospective control group not receiving meals at two other KPCO-contracted hospitals.

Hypothesis 3: Patients receiving meals for 4 weeks will have a decreased composite rate of rehospitalizations and ED visits at 60 days compared to those receiving meals for 2 weeks or the non-randomized control group.

Specific Aim 4: To determine the feasibility, acceptability and scalability of the Meals Matter Program to KP members, their households, and hospital leadership and staff.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older, with no upper age limit
* Hospitalized at Saint Joseph Hospital or Good Samaritan Medical Center with the anticipation that they will be discharged home
* Member of a KP health plan
* Have one or more of the following conditions:

  * Heart failure
  * Cancer
  * End-stage renal disease (ESRD)/chronic renal disease
  * Chronic obstructive pulmonary disease (COPD)
  * Diabetes Mellitus
  * Chronic liver disease/cirrhosis

Exclusion Criteria:

* Patient discharged to a nursing home, an assisted living facility, or another setting where meals are institutionally provided
* Patient has a health condition which is incompatible with the diet choices offered by Project Angel Heart (PAH - food service vendor)
* Patient refuses the type of meal best for their medical condition
* Patient has dementia
* Patient is pregnant or hospitalized peri-partum
* Patient is an active participant in a PAH program or another meal program
* Patient is unable to speak English or Spanish
* PAH unable to deliver meals due to patient not being in PAH service area
* Patient was discharged from the hospital within 24 hours of admission
* Patient whose household member has enrolled in the Meals MATTER study
* Patient discharged to hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Anxiety and Depression measured through the Hospital Anxiety and Depression Scale | A change in score from baseline to 60 days
  Measured through the Hospital Anxiety and Depression Scale. 0 = Minimum. 21 = Maximum. Higher score is worse outcome.

SECONDARY OUTCOMES:
Functional Status measured through the Katz Activities of Daily Living Scale | A change in score from baseline to 60 days
  Measured through the Katz Activities of Daily Living. Minimum = 0, Maximum = 6. Higher score is better outcome.
Re-hospitalization and Emergency Department Visits | 60 days from hospital discharge
  Measured through time of discharge through re-hospitalization or Emergency Department visit

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S Boxer, MD, MS, Principal Investigator — KP Institute for Health Research; John Steiner, MD, MPH, Study Director — KP Institute for Health Research
Locations (2):
- United States (2):
  - St Joseph's Hospital, Denver, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado